CLINICAL TRIAL: NCT02217722
Title: An Open Label Non Randomized Pilot Study: Use of the Ulcerative Colitis Diet for Induction of Remission.
Brief Title: Use of the Ulcerative Colitis Diet for Induction of Remission
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We have submitted a multi center study, with the same nutritional therapy
Sponsor: Prof. Arie Levine (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition unit., Wolfson Medical Center
Organization: Wolfson Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0096-14-WOMC
Record Dates: First submitted 2014-07-20; First posted 2014-08-15 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Doxycycline; Amoxicillin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ulcerative Colitis Diet counseling (Experimental): Patients will receive a structured novel diet termed the UCD for 6 weeks. . patients that completed induction phase with remission(PUCAI<10) will be asked if they are willing to adhere to the UCD for an additional 20 weeks.
  Interventions: Other: Ulcerative Colitis Diet
- Antibiotic Treatment (Experimental): Patients failing to enter or maintain remission by 6 weeks, or with worsening disease at any time after week 2 will be considered failures on an intention to treat basis. Eligible patients at this time at aged 10 or above may receive a 14 day antibiotic course with Doxycycline, amoxicillin and metronidazole.In addition to the description above children who refused to UCD or with low adherence to UCD may be enrolled directly to this arm.
  Interventions: Drug: Antibiotic cocktail

INTERVENTIONS:
Other: Ulcerative Colitis Diet — we have postulated that a diet that increases butyrate through fiber exposure, reduces intestinal sulfur exposure, and increases vitamin D levels could be beneficial for patients with Ulcerative Colitis. To date, no study has explored this possibility.
  Arms: Ulcerative Colitis Diet counseling
Drug: Antibiotic cocktail — We have postulating that antibiotic therapy can alter the microbiota clinically. Controlling the microbiota by antibiotics may allow for control of the disease without immune suppression
  Other Names: Doxycyclin, amoxicillin and metronidazole
  Arms: Antibiotic Treatment

SUMMARY:
The goal of the study is to evaluate the use of Ulcerative Colitis Diet for Induction of Remission. The investigators have postulated that we developed could be beneficial for patients with Ulcerative Colitis. To date, no study has explored this possibility.

DETAILED DESCRIPTION:
Background:

Recent research has shown that dietary components may lead to impaired intestinal innate immunity due to alterations in the microbiome, mucous layer, intestinal permeability or change in bacterial adherence and translocation. Pfeffer Gik et al (Dig Dis, 2014) compiled a list of food components and additives that impair the intestinal epitheliums ability to contain bacteria to the lumen, and consequently increase intestinal permeability which, in turn, increases the uptake of luminal antigens and microbial factors. The list includes Gliadin, Saturated fat milks, emulsifiers such as Carboxymethylcellulose, Polysorbate 80 and Sodium Caprate )Levine A, Wine E, 2013). In Crohn's disease, intervention with EEN or a Crohn's disease exclusion diet have shown high rates of remission in mild- moderate CD patients. The CDED led to remission in 70% of patients, primarily with patients with early mild to moderate disease (Sigall-Boneh R et al, 2014).

Unlike CD, none of these studies have systematically examined the relationship between normal diet intake and relapses in UC. Devotka et al demonstrated that a bloom in sulphide reducing bacteria increased colitis in IL10-/- mice. This was due to increased Bilophila Wadsworthia which is sulphide dependent (Brown k et al, 2012). Studies have shown that the rate of butyrate utilization in normal specimens was almost double than that found in UC Specimens. Moreover, high fiber diet can affect the microbial composition (Pitcher MCL et al, Gut, 2000) and regulatory T cells in the colon (Singh N et al, 2014).

Until recently, UC was not considered to be a bacteria mediated disease. However, our increased understanding of UC indicates that bacteria might have a role in pathogenesis or severity of the disease. The strongest evidence comes from Japanese studies in patients with moderate to severe colitis, which demonstrated that triple therapy with penicillin , tetracycline and metronidazole led to remission in steroid refractory patients in 60% of patients, and this was reproduced in a follow up randomized controlled trial which showed a 70% remission rate (UEGW Amsterdam 2012, Ohkusa T et al 2005 ). On the other hand a previous trial had shown 44% response and only (Ohkusa T et al 2010). A recent retrospective study in Israel showed a 65% response and 50% remission rate in patients with severe refractory colitis. Thus it is unclear at present if antibiotics are useful only in severe colitis , or if this reflects heterogeneity among studies.

Diet and antibiotics are the two proven treatments that may alter the microbiota clinically. Theoretically, controlling the microbiota by diet or antibiotics may allow for control of the disease without immune suppression , and this has yet to be evaluated.

Based on our previous success in improving remission and decreasing inflammation with a novel dietary intervention in Crohn's disease, and based on these previously mentioned studies, we have postulated that a diet could be beneficial for patients with Ulcerative Colitis. We further hypothesize that patients failing diet might respond to antibiotic therapy If patients respond to the diet this would have an immediate impact and be the first evidence for a specific diet that works in UC. If the diet fails and the antibiotics succeed, this would be the first evidence for the effect of oral antibiotics in mild disease .

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Established diagnosis of UC disease.
* Age: 5 - 18 years ( inclusive)
* Mild to moderate active disease, 10 ≤ PUCAI ≤45.
* Stable medication (IMM/ 5ASA) use for the past 6 weeks.
* For patients who received antibiotic treatment: age 10-18 (inclusive).

Exclusion Criteria:

* Any proven infection such as positive stool culture, parasite or C.difficile.
* Use of Antibiotics
* Use of steroids in the previous two weeks only
* Patients that are refractory to full dose steroids ( 1 mg/kg/day)
* Past acute severe UC.
* Current Extra intestinal manifestation of UC.
* Pregnancy.

A subset of patients who are on steroids and relapse during steroids treatment ≤0.5 mg/kg with mild to moderate disease activity will act as a second subset for this exploratory study.

-

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Remission rate, defined as a PUCAI less than 10 at week 6. | week 6

SECONDARY OUTCOMES:
Change in Mean PUCAI week 6. | week 6
Change in mean Calprotectin week 6 | week 6

CONTACTS AND LOCATIONS:
Locations (1):
- The E.Wolfson Medical Center, Holon, Israel